CLINICAL TRIAL: NCT03637504
Title: Feasibility of a Mobile Medication Plan Application in CF Patient Care
Acronym: MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of Arizona (Other); Johns Hopkins University (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Gregory Sawicki, Co-Chair of Success with Therapies Research Consortium, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00021541; STRC-102-17-01 (Other: Success with Therapies Research Consortium)
Record Dates: First submitted 2018-07-26; First posted 2018-08-20 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis in Children
Keywords: Feasibility; Mobile Medication Plan Application; Patient Care; Nebulized Medications; Oral Medications; MedActionPlan; eTrack Nebulizer; AdhereTech Pill Bottles
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interventional (Experimental): web-based, mobile medication management application [MedActionPlan® (MAP) and continued use of eTrack nebulizer +/- AdhereTech pill bottles as measures of adherence
  Interventions: Behavioral: MedActionPlan®
- Control (No Intervention): usual care and continued use of eTrack nebulizer +/- AdhereTech pill bottles as measures of adherence
- Optional Extension (Other): web-based, mobile medication management application [MedActionPlan® (MAP)]
  Interventions: Behavioral: MedActionPlan®

INTERVENTIONS:
Behavioral: MedActionPlan® — web-based, mobile medication management application [MedActionPlan® (MAP)]
  Other Names: MAP
  Arms: Interventional; Optional Extension

SUMMARY:
This is a pilot, multicenter, prospective, randomized controlled study to evaluate the feasibility of an innovative medication adherence intervention utilizing a web-based, mobile medication management application [MedActionPlan® (MAP)] to encourage self-management by reinforcing adherence and education about treatment regimens in Participants with cystic fibrosis (CF) (ages 12 years and older).

Outcomes of interest for this study are 1) feasibility of MAP in real-world setting which will be evaluated using patient/caregiver and clinician feedback regarding value, ease of use, and challenges with use, 2) effect of MAP on patient/caregiver knowledge and perception of medication use, 3) effect of MAP on adherence to inhaled and oral medications used in chronic management of CF. Preliminary data regarding outcomes on exacerbations, lung function, and health care system utilization (e.g., emergency department visits, hospitalization) will also be examined as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* CLINICIAN PARTICIPANTS:

  1. A CF care team member from any discipline, designated by the site principal investigator (PI) and CF team
  2. Willing to use MAP as part of CF care
* PATIENT PARTICIPANTS:

  1. Male or female patients ages ≥ 12 years of age at Study Visit 1
  2. Documentation of a CF diagnosis (physician diagnosed)
  3. Ability to understand verbal and written English
  4. Access to mobile device such as a tablet or smartphone (iPhone/iPad/iTouch or Android device)
  5. Willingness to use the MAP application
  6. Currently taking at least one of the following chronic medications and willing to use AdhereTech pill bottles for oral medications and/or eTrack nebulizer for nebulized medications listed below: nebulized agents, dornase alfa, hypertonic saline, inhaled tobramycin, inhaled aztreonam, inhaled colistimethate, oral agents, azithromycin
* CAREGIVER PARTICIPANTS (for Patient Participants age < 18 years)

  1. Child is consented to participate in the study.
  2. Ability to understand verbal and written English

Exclusion Criteria:

* CLINICIAN PARTICIPANTS:

Previous use of MAP (with patient(s) or self) in the last 12 months - when used with patients, defined as use in 5 or more patients

* PATIENT PARTICIPANTS:

  1. Previous use of MAP in the last 12 months - defined as use for 4 weeks or longer in own care
  2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data including, but not limited to, diagnosis of intellectual or developmental disability (e.g., autism); and/or history of lung transplant
  3. Planned or scheduled hospitalization during study period of up to 36 weeks
* CAREGIVER PARTICIPANTS:

(for Patient Participants age < 18 years)

1. Previous use of MAP in the last 12 months - defined as use for 4 weeks or longer in child's or own care

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
mean score of Intervention Feasibility and Acceptability questionnaire (iFAQ) for patients assessed by likert scale | week 24
  This measure was developed for this specific study to evaluate feasibility and acceptability of patient use through aspects of usability and quality (engagement, usefulness, functionality/ease of use, aesthetics, information, and satisfaction) of the web portal and application. Assessed by 5 point Likert Scale: Strongly disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree
mean score of Intervention Feasibility and Acceptability questionnaire (iFAQ) for clinicians assessed by likert scale | up to 30 months
  This measure was developed for this specific study to evaluate feasibility and acceptability of clinician use through aspects of usability and quality (engagement, usefulness, functionality/ease of use, aesthetics, information, and satisfaction) of the web portal and application. Assessed by 5 point Likert Scale: Strongly disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree

SECONDARY OUTCOMES:
change in Knowledge of Disease Management-CF questionnaire (KDM-CF) scores | Day 1 to approximately week 24
  This validated measure was developed for studies of adherence and disease management. It assesses the practical knowledge of patients with CF. The measure evaluates knowledge of disease management in four areas (general health, lung health, nutrition, treatments).Data regarding changes in knowledge (using KDM-CF), from baseline to end of study visit, will be analyzed using Wilcoxon Signed Rank test. Data regarding changes in knowledge (using KDM-CF and CF-MQ) between groups (Intervention vs. Control) will be analyzed using Wilcoxon Rank Sum test.
change in CF Medication Belief Questionnaire (CF-MBQ) scores | Day 1 to approximately week 24
  Developed and validated to measure impact of interventions on specific social cognitive beliefs. Data regarding perception of medications (using CF-MBQ), from baseline to end of study, will be analyzed using Wilcoxon Signed Rank test. Data regarding perception of medications (using CF-MBQ), between groups (Intervention vs. Control), will be analyzed using Wilcoxon Rank Sum test. The CF-MBQ has 60 questions. There are five domains for this measure: motivation, self-efficacy, perceived importance of medication, and decisional balance to take or miss medications. Questions related to self-efficacy, motivation and importance items use a scale from 1 to 10. Questions related to decisional balance use a scale based on a 1 to 5 scale. Scores for each subscale's items will be summed and divided by the number of items to produce an average score ranging from 1 to 10 (self-efficacy, motivation and importance) OR 1 to 5 (decisional balance).
Mean change in adherence | Day 1 to approximately week 24
  Assess the preliminary effect of MAP on medication adherence from data collected from AdhereTech pill bottles and eTrack nebulizers that will be scored as a 'per drug analysis' of adherence with a ratio of competed to total prescribed doses in the study period. A composite score will be determined based on prescribed medications and medication/doses taken.
change in CF Medication Questionnaire (CF-MQ) scores | Day 1 to approximately week 24
  Developed to assess Patient Participant knowledge about prescribed CF medications including purpose, dose, and administration. Question items will evaluate knowledge of medication purpose, administration, dose, and dosing frequency. Correct response for dose and dosing frequency will be based on each patient's prescribed regimen. Questions regarding medication purposes and appropriate administration each have 1 correct answer. Total score will be defined as proportion of correct items to total items asked. Each Patient Participant will only be asked about items that are associated with that Patient Participant's prescribed treatment plan. Total score for a Participant will not be calculated if greater than 20% of the items are missing responses.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Phan, Principal Investigator — University of Michigan; Cori Daines, Principal Investigator — University of Arizona
Locations (5):
- United States (5):
  - Children's of Alabama, Birmingham, Alabama
  - University of Arizona and Banner Health, Tucson, Arizona
  - Lucille Packard Children's Hospital Stanford, Stanford, California
  - Johns Hopkins University, Baltimore, Maryland
  - University at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No